CLINICAL TRIAL: NCT02965859
Title: A Randomized,Double-blind,Double-dummy,Multiple-dose Parallel Control,Multiple Centers Study to Assess the Safety and Dose-range of Metacavir Enteric-coated Capsules for Patients With Chronic Hepatitis B
Brief Title: The Safety and Dose-range Study of Metacavir Enteric-coated Capsules in Patients With Chronic Hepatitis B
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Yipinhong Pharmaceutical CO.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNA-20140110-v2
Record Dates: First submitted 2016-09-01; First posted 2016-11-17 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir dipivoxil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Metacavir Enteric-coated Capsule 80mg (Experimental): 1. Metacavir Enteric-coated Capsules 80mg
  2. Metacavir Enteric-coated Capsules Placebo 240mg
  3. Adefovir Dipivoxil Capsule Placebo 10mg;
  Interventions: Drug: Metacavir Enteric-coated Capsules 80mg; Drug: Metacavir Enteric-coated Capsules Placebo 240mg; Drug: Adefovir Dipivoxil Capsule Placebo 10mg
- Metacavir Enteric-coated Capsules 160mg (Active Comparator): 1. Metacavir Enteric-coated Capsules 160mg
  2. Metacavir Enteric-coated Capsules Placebo 160mg
  3. Adefovir Dipivoxil Capsule Placebo 10mg;
  Interventions: Drug: Metacavir Enteric-coated Capsules 160mg; Drug: Metacavir Enteric-coated Capsules Placebo 160mg; Drug: Adefovir Dipivoxil Capsule Placebo 10mg
- Metacavir Enteric-coated Capsules 320mg (Placebo Comparator): 1. Metacavir Enteric-coated Capsules 320mg
  2. Adefovir Dipivoxil Capsule Placebo 10mg
  Interventions: Drug: Metacavir Enteric-coated Capsules 320mg; Drug: Adefovir Dipivoxil Capsule Placebo 10mg
- Adefovir Dipivoxil Capsule (Active Comparator): 1. Metacavir Enteric-coated Capsules Placebo 320mg
  2. Adefovir Dipivoxil Capsule 10mg;
  Interventions: Drug: Metacavir Enteric-coated Capsules Placebo 320mg; Drug: Adefovir Dipivoxil Capsule10mg
- Placebo (Placebo Comparator): 1. Metacavir Enteric-coated Capsules Placebo 320mg
  2. Adefovir Dipivoxil Capsule Placebo 10mg;
  Interventions: Drug: Metacavir Enteric-coated Capsules 320mg; Drug: Metacavir Enteric-coated Capsules Placebo 320mg; Drug: Adefovir Dipivoxil Capsule Placebo 10mg

INTERVENTIONS:
Drug: Metacavir Enteric-coated Capsules 80mg — Metacavir Enteric-coated Capsules 80mg
  Arms: Metacavir Enteric-coated Capsule 80mg
Drug: Metacavir Enteric-coated Capsules 160mg — Metacavir Enteric-coated Capsules 160mg
  Arms: Metacavir Enteric-coated Capsules 160mg
Drug: Metacavir Enteric-coated Capsules 320mg — Metacavir Enteric-coated Capsules 320mg
  Arms: Metacavir Enteric-coated Capsules 320mg; Placebo
Drug: Metacavir Enteric-coated Capsules Placebo 240mg — Metacavir Enteric-coated Capsules Placebo 240mg
  Arms: Metacavir Enteric-coated Capsule 80mg
Drug: Metacavir Enteric-coated Capsules Placebo 160mg — Metacavir Enteric-coated Capsules Placebo 160mg
  Arms: Metacavir Enteric-coated Capsules 160mg
Drug: Metacavir Enteric-coated Capsules Placebo 320mg — Metacavir Enteric-coated Capsules Placebo 320mg
  Arms: Adefovir Dipivoxil Capsule; Placebo
Drug: Adefovir Dipivoxil Capsule10mg — Adefovir Dipivoxil Capsule10mg
  Arms: Adefovir Dipivoxil Capsule
Drug: Adefovir Dipivoxil Capsule Placebo 10mg — Adefovir Dipivoxil Capsule Placebo 10mg
  Arms: Metacavir Enteric-coated Capsule 80mg; Metacavir Enteric-coated Capsules 160mg; Metacavir Enteric-coated Capsules 320mg; Placebo

SUMMARY:
The study objective is to evaluate the safety and effectiveness of different doses of Metacavir Enteric-coated Capsules in treatment of chronic hepatitis B,as well as to find an appropriate clinical dosage by comparing the effect of different doses of treatment,in order to provide references of clinical trial of the next phase.

DETAILED DESCRIPTION:
180 eligible subjects will be included.According to the set grouping method of dose escalation.Subjects will be randomized in a 1:1:1:1 proportion of Metacavir Enteric-coated Capsules(80mg/160mg/320mg) group,positive control group or placebo control group.Each group has 36 subjects.

1.Subjects will use the study medication(2 hours before or after meal,once a day) from Visit 3 to Visit 5.

1. Metacavir Enteric-coated Capsules 80mg Group:Metacavir Enteric-coated Capsules 80mg,Metacavir Enteric-coated Capsules Placebo 240mg,Adefovir Dipivoxil Capsule Placebo 10mg;
2. Metacavir Enteric-coated Capsules 160mg Group:Metacavir Enteric-coated Capsules 160mg,Metacavir Enteric-coated Capsules Placebo 160mg,Adefovir Dipivoxil Capsule Placebo 10mg;
3. Metacavir Enteric-coated Capsules 320mg Group:Metacavir Enteric-coated Capsules 320mg,Adefovir Dipivoxil Capsule Placebo 10mg;
4. Positive Control(Adefovir Dipivoxil Capsule) Group:Metacavir Enteric-coated Capsules Placebo 320mg,Adefovir Dipivoxil Capsule 10mg;
5. Placebo Control Group:Metacavir Enteric-coated Capsules Placebo 320mg,Adefovir Dipivoxil Capsule Placebo 10mg;

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age and no older than 65;
* Subjects,with an established clinical history of HBV at Screening,has a positive HBsAg test(>6months) regardless of a positive/negative HBeAg test;
* At Screening,HBV-DNA>10^5 copies/ml in HBeAg positive or HBV-DNA>10^4 copies/ml in HBeAg negative(HBV-DNA was evaluated by polymerase chain reaction fluorescent labeling.);
* Subjects with abnormal liver function test defined as alanine aminotransferase(ALT) was 2~10 times upper limit of normal in HBeAg positive or 1.5~10 times upper limit of normal in HBeAg negative;
* Subjects who are willing to require any other treatment for anti-hepatitis B during the study period;
* Subjects who are willing to take measures for effective non-pharmaceutical contraception;
* Given their signed written informed consent to participate;

Exclusion Criteria:

* Subjects with hepatitis C(HCV),hepatitis D(HDV),autoimmune hepatitis,hereditary liver disease or any other active hepatitis;
* A positive human immunodeficiency virus(HIV) test result;
* Subjects,who in the opinion of the investigator,have a current diagnosis of hepatocellular carcinoma or serum α-fetoprotein(AFP)>100ug/L;
* Subjects with severe hepatitis or decompensated liver disease defined as hepatic encephalopathy,ascites,low protein blood syndrome(albumin ≤30g/l) or variceal bleeding;
* Serum Creatinine(SCr) exceeds upper limit of normal;
* At Screening,ALT>10 times upper limit of normal,Total Bilirubin(TBIL)>double upper limit of normal or transient hepatic decompensation caused by condition aggravation;
* Subjects who required treatment with nucleoside antiviral drugs such as lamivudine,Adefovir dipivoxil,Telbivudine,Tenofovir disoproxil or Entecavir before Screening;
* Subjects who require treatment with interferon-α，thymosin α-1 or other antiviral therapy,immunosuppressive agents,immune modulators within 6 months before Screening;
* Subjects with cardiac disease,hematological system disease,cancer,impaired immunity or psychiatric disease;
* Hemoglobin<10g/dl,white blood cell count<3.5 10^9/L,platelets<80 10^9/L;
* Subjects,who in the opinion of the investigator,have a current diagnosis of pancreatitis pre-dose within 24 weeks;
* History of hypersensitivity or allergy to any of the study drugs;
* Subjects who participate in other clinical trials within 3 months prior to Screening;
* Women who are pregnant or lactating or planning a pregnancy recently;
* Subjects in the opinion of the investigator,could not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the logarithms of measurement data of HBV-DNA at Week 12 of treatment. | 12 weeks
  The change from baseline in the logarithms of measurement data of HBV-DNA at Week 12 of treatment.（Unit：log10)

SECONDARY OUTCOMES:
Incidence of treatment-chronic hepatitis B | 12 weeks
  1. The proportion of subjects whose HBV-DNA are down to double logarithms at Week 12 of treatment.(Unit：%)
  2. The proportion of subjects whose HBV-DNA are not detected or less than upper limit of normal at Week 12 of treatment.(Unit：%)
  3. The proportion of subjects (HBeAg positive at baseline) whose is changed at Week 12 of treatment.(Unit：%)
  4. The proportion of subjects whose HBsAg is changed to negative at Week 12 of treatment.(Unit：%)
Incidence of Adverse Events(AEs) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maorong Wang, Principal Investigator — 81 Military Hospital of China; Yonggang Li, Principal Investigator — Beijing 302 Hospital; Yongfeng Yang, Principal Investigator — The Second Hospital of Nanjing Medical University; Yanlin Yu, Principal Investigator — Wannan Medical College Yijishan Hospital; Jun Li, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- 81 Military Hospital of China, Nanjing, Jiangsu, China